CLINICAL TRIAL: NCT04602221
Title: A Randomized, Placebo Controlled, Double-blind, Double-dummy Three-way Cross Over Trial to Investigate the Effect of BI 409306, BI 425809 and Lamotrigine on Ketamine-induced Cognitive Deficits in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test Whether BI 409306, BI 425809 or Lamotrigine Can Reverse the Memory Problems Caused by Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1289-0057
Record Dates: First submitted 2020-10-16; First posted 2020-10-26 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Lamotrigine; BI 409306; BI 425809

STUDY DESIGN:
Intervention Model Description: 3-treatment period design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Treatment sequence: T1-T2-R (Experimental): Treatments:
  T1: Lamotrigine T2: BI 409306 T3: BI 425809 R: Placebo
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: T1-R-T2 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: T1-T3-R (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T1-R-T3 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T2-T1-R (Experimental)
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: T2-R-T1 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: T2-T3-R (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T2-R-T3 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T3-R-T1 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T3-T1-R (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T3-T2-R (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809
- Treatment sequence: T3-R-T2 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809
- Treatment sequence: R-T1-T2 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: R-T2-T1 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: BI 409306; Drug: Placebo
- Treatment sequence: R-T1-T3 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: R-T3-T1 (Experimental)
  Interventions: Drug: Lamotrigine; Drug: Placebo; Drug: BI 425809
- Treatment sequence: R-T2-T3 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809
- Treatment sequence: R-T3-T2 (Experimental)
  Interventions: Drug: BI 409306; Drug: Placebo; Drug: BI 425809

INTERVENTIONS:
Drug: Lamotrigine — Tablet
  Arms: Treatment sequence: R-T1-T2; Treatment sequence: R-T1-T3; Treatment sequence: R-T2-T1; Treatment sequence: R-T3-T1; Treatment sequence: T1-R-T2; Treatment sequence: T1-R-T3; Treatment sequence: T1-T2-R; Treatment sequence: T1-T3-R; Treatment sequence: T2-R-T1; Treatment sequence: T2-T1-R; Treatment sequence: T3-R-T1; Treatment sequence: T3-T1-R
Drug: BI 409306 — Film-coated tablet
  Arms: Treatment sequence: R-T1-T2; Treatment sequence: R-T2-T1; Treatment sequence: R-T2-T3; Treatment sequence: R-T3-T2; Treatment sequence: T1-R-T2; Treatment sequence: T1-T2-R; Treatment sequence: T2-R-T1; Treatment sequence: T2-R-T3; Treatment sequence: T2-T1-R; Treatment sequence: T2-T3-R; Treatment sequence: T3-R-T2; Treatment sequence: T3-T2-R
Drug: Placebo — Tablet, Film-coated tablet
Drug: BI 425809 — Film-coated tablet
  Arms: Treatment sequence: R-T1-T3; Treatment sequence: R-T2-T3; Treatment sequence: R-T3-T1; Treatment sequence: R-T3-T2; Treatment sequence: T1-R-T3; Treatment sequence: T1-T3-R; Treatment sequence: T2-R-T3; Treatment sequence: T2-T3-R; Treatment sequence: T3-R-T1; Treatment sequence: T3-R-T2; Treatment sequence: T3-T1-R; Treatment sequence: T3-T2-R

SUMMARY:
The main objective of this trail is to investigate if and to what extent BI 409306, BI 425809 and lamotrigine attenuate ketamine induced cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. BMI of 18.5 to 32 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
5. Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

   * Use of adequate contraception, e.g. use of condom (male subjects) plus any of the following methods (female partners): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide)
   * Sexually abstinent
   * Vasectomised (vasectomy at least 1 year prior to enrolment)
   * Surgically sterilised female partner (including hysterectomy, bilateral tubal occlusion or bilateral oophorectomy)
   * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea

Exclusion Criteria:

1. Any finding in the medical examination (including ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. History of diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical trial was performed as a randomised, placebo-controlled, double-blind, doubledummy, three-way crossover trial in healthy male subjects to investigate if and to what extent BI 409306, BI 425809, and lamotrigine attenuated ketamine-induced cognitive deficits
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Treatment Sequence: R-T3-T2: Subjects randomized to treatment sequence R-T3-T2 received reference treatment R in period 1, test treatment T3 in period 2 and test treatment T2 in period. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of Placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride were administered intravenously at 5:00 hours (planned time).
  Treatment periods was separated by a washout period of at least 11 days.
- Treatment Sequence: R-T3-T1: Subjects randomized to treatment sequence R-T3-T1 received reference treatment R in period 1, test treatment T3 in period 2 and test treatment T1 in period 3. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of Placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: R-T2-T3: Subjects randomized to treatment sequence R-T2-T3 received reference treatment R in period 1, test treatment T2 in period 2 and test treatment T3 in period 3. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of Placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: R-T2-T1: Subjects randomized to treatment sequence R-T2-T1 received reference treatment R in period 1, test treatment T2 in period 2 and test treatment T1 in period 3. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of Placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: R-T1-T3: Subjects randomized to treatment sequence R-T1-T3 received reference treatment R in period 1, test treatment T1 in period 2 and test treatment T3 in period 3. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: R-T1-T2: Subjects randomized to treatment sequence R-T1-T2 received reference treatment R in period 1, test treatment T1 in period 2 and test treatment T2 in period 3. Treatments were administered on Day 1 of each treatment period.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T3-R-T2: Subjects randomized to treatment sequence T3-R-T2 received test treatment T3 in period 1, reference treatment R in period 2 and test treatment T2 in period 3. Treatments were administered on Day 1 of each treatment period.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T3-R-T1: Subjects randomized to treatment sequence T3-R-T1 received test treatment T3 in period 1, reference treatment R in period 2 and test treatment T1 in period 3. Treatments were administered on Day 1 of each treatment period.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T3-T2-R: Subjects randomized to treatment sequence T3-T2-R received test treatment T3 in period 1, test treatment T2 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T3-T1-R: Subjects randomized to treatment sequence T3-T1-R received test treatment T3 in period 1, test treatment T1 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T2-R-T3: Subjects randomized to treatment sequence T2-R-T3 received test treatment T2 in period 1, reference treatment R in period 2 and test treatment T3 in period 3. Treatments were administered on Day 1 of each treatment period.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T2-R-T1: Subjects randomized to treatment sequence T2-R-T1 received test treatment T2 in period 1, reference treatment R in period 2 and test treatment T1 in period 3. Treatments were administered on Day 1 of each treatment period.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T2-T3-R: Subjects randomized to treatment sequence T2-T3-R received test treatment T2 in period 1, test treatment T3 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T2-T1-R: Subjects randomized to treatment sequence T2-T1-R received test treatment T2 in period 1, test treatment T1 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T1-R-T3: Subjects randomized to treatment sequence T1-R-T3 received test treatment T1 in period 1, reference treatment R in period 2 and test treatment T3 in period 3. Treatments were administered on Day 1 of each treatment period.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T1-R-T2: Subjects randomized to treatment sequence T1-R-T2 received test treatment T1 in period 1, reference treatment R in period 2 and test treatment T2 in period 3. Treatments were administered on Day 1 of each treatment period.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T1-T3-R: Subjects randomized to treatment sequence T1-T3-R received test treatment T1 in period 1, test treatment T3 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose.
  At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  T3: At 0:00 hours (planned time): one film-coated tablet of 25 mg BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of placebo to BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
- Treatment Sequence: T1-T2-R: Subjects randomized to treatment sequence T1-T2-R received test treatment T1 in period 1, test treatment T2 in period 2 and reference treatment R in period 3. Treatments were administered on Day 1 of each treatment period.
  T1: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): three tablets of 100 mg Lamotrigine and one film-coated tablet of placebo to BI 409306 as single oral dose each.
  T2: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809, as single oral dose. At 03:00 hours (planned time): one film-coated tablet of 50 mg BI 409306 and three film coated tablets of placebo to lamotrigine, as single oral dose each.
  R: At 00:00 hours (planned time): one film-coated tablet of placebo to BI 425809 as single oral dose. At 03:00 hours (planned time): three film-coated tablets of placebo to lamotrigine and one film-coated tablet of placebo to BI 409306, as single oral dose each.
  In each treatment period 500 mg/10 milliliter solution for injection of Ketamine hydrochloride was administered intravenously at 5:00 hours (planned time). Treatment periods were separated by a washout period of at least 11 days.
Period: Overall Study
Arm/Group | Treatment Sequence: R-T3-T2 | Treatment Sequence: R-T3-T1 | Treatment Sequence: R-T2-T3 | Treatment Sequence: R-T2-T1 | Treatment Sequence: R-T1-T3 | Treatment Sequence: R-T1-T2 | Treatment Sequence: T3-R-T2 | Treatment Sequence: T3-R-T1 | Treatment Sequence: T3-T2-R | Treatment Sequence: T3-T1-R | Treatment Sequence: T2-R-T3 | Treatment Sequence: T2-R-T1 | Treatment Sequence: T2-T3-R | Treatment Sequence: T2-T1-R | Treatment Sequence: T1-R-T3 | Treatment Sequence: T1-R-T2 | Treatment Sequence: T1-T3-R | Treatment Sequence: T1-T2-R
Started | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Discontinuation of trial treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other than listed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were randomised and treated with at least one dose of Investigational medicinal product (IMP)/Placebo or ketamine.
Groups:
- Total: All participants that were treated with at least one dose of Investigational medicinal product (IMP)/Placebo or ketamine.
Arm/Group | Total
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 17
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Paired Associate Learning (PAL) Total Errors Adjusted (PALTEA28) on Ketamine
Description: Paired Associate Learning (PAL) assesses visual memory and new learning. Boxes are displayed on the screen and open in turn to reveal a number of patterns. Participants are instructed to try to remember the location in which each pattern was shown. After all the boxes have been opened, each pattern is then shown in the center of the screen in a randomised order, and the participant touches the box in which the pattern was located. If an error is made, all the patterns are re-presented to remind the participant of their locations.
  The PALTEA28 evaluates the number of errors committed by the subject plus an adjustment for the estimated number of errors they would have made on any stages that were not reached. Calculated across all assessed two, four, six and eight box trials.
Time Frame: At 4:20 and 5:06 hours:minutes after first drug administration in each treatment period.
Population: Pharmacodynamic (PD) set (PDS): PD analyses were based on the PDS which was defined as all randomised subjects who performed the post ketamine tests in at least one period. Number of participants differs due to incomplete crossover design.
Measure: Least Squares Mean (Standard Error); unit: Errors
Groups:
- Placebo (R): One film-coated tablet of Placebo to BI 409306 and three film-coated tablets of placebo to lamotrigine were administered as oral single dose each, 2 hours prior to ketamine infusion on Day 1 and one film-coated tablet of Placebo to BI 425809 was administered as oral single dose 5 hours prior to ketamine infusion on Day 1.
- 25 mg BI 425809 (T3): 1 film-coated tablet of 25 milligrams (mg) BI 425809 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T3, 5 hours prior to ketamine infusion.
- 50 mg BI 409306 (T2): 1 film-coated tablet of 50 milligrams (mg) BI 409306 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T2, 2 hours prior to ketamine infusion.
- 300 mg Lamotrigine (T1): 3 tablets of 100 milligrams (mg) Lamotrigine were administered orally once daily (daily dose: 300 mg) with 240 mL of water after a light snack on Day 1 of treatment T1, 2 hours prior to ketamine infusion.
Arm/Group | Placebo (R) | 25 mg BI 425809 (T3) | 50 mg BI 409306 (T2) | 300 mg Lamotrigine (T1)
Number analyzed (Participants) | 34 | 23 | 23 | 26
Errors | 24.169 (2.5972) | 23.829 (3.2275) | 28.170 (3.2334) | 22.911 (3.0850)
Statistical Analysis 1: Comparison: Placebo (R) vs 25 mg BI 425809 (T3); A linear mixed effects model, i.e. analyses of covariance (ANCOVA) was used for analysis of the primary endpoint. This model included effects for sequence, subject within sequence, period, baseline values (pre-ketamine baseline and on-ketamine baseline) and treatment. The effect 'subject within sequence' were considered as random, whereas the other effects were considered as fixed; Test type: Other; p = 0.9296, ANCOVA; Difference of adjusted means = -0.339, 95% CI 2-sided [-7.975 to 7.297], Standard Error of Mean 3.8242 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 2: Comparison: Placebo (R) vs 50 mg BI 409306 (T2); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2990, ANCOVA; Difference of adjusted means = 4.002, 95% CI 2-sided [-3.631 to 11.634], Standard Error of Mean 3.8224 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 3: Comparison: Placebo (R) vs 300 mg Lamotrigine (T1); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7322, ANCOVA; Difference of adjusted means = -1.258, 95% CI 2-sided [-8.565 to 6.050], Standard Error of Mean 3.6608 — The difference was calculated as treatment group minus placebo group

2. Secondary Outcome: Spatial Working Memory (SWM) Between Errors (BE468) on Ketamine
Description: SWM assesses the ability of the participant to retain spatial information and manipulate it in working memory. A number of coloured boxes are presented on the screen, and the computer hides a token in these boxes one at a time. The participant is instructed to touch the boxes in turn to search for the token that has been hidden. The key task instruction is that the computer will never hide a token in the same coloured box twice in the same problem.
  The SWMBE468 evaluates the number of times the subject incorrectly revisits a box in which a token has previously been found. Calculated across all assessed four, six and eight token trials.
Time Frame: At 4:20 and 5:06 hours:minutes after first drug administration in each treatment period.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Errors
Groups:
- 25mg BI 425809 (T3): 1 film-coated tablet of 25 milligrams (mg) BI 425809 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T3, 5 hours prior to ketamine infusion.
- 50mg BI 409306 (T2): 1 film-coated tablet of 50 milligrams (mg) BI 409306 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T2, 2 hours prior to ketamine infusion.
Arm/Group | Placebo (R) | 25mg BI 425809 (T3) | 50mg BI 409306 (T2) | 300 mg Lamotrigine (T1)
Number analyzed (Participants) | 33 | 23 | 22 | 25
Errors | 15.684 (1.3412) | 16.032 (1.5427) | 14.600 (1.5704) | 12.826 (1.5005)
Statistical Analysis 1: Comparison: Placebo (R) vs 25mg BI 425809 (T3); A linear mixed effects model, i.e. analyses of covariance (ANCOVA) was used for analysis of the secondary endpoint. This model included effects for sequence, subject within sequence, period, baseline values (pre-ketamine baseline and on-ketamine baseline) and treatment. The effect 'subject within sequence' were considered as random, whereas the other effects were considered as fixed; Test type: Other; p = 0.8249, ANCOVA; Difference of adjusted means = 0.347, 95% CI 2-sided [-2.776 to 3.471], Standard Error of Mean 1.5630 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 2: Comparison: Placebo (R) vs 50mg BI 409306 (T2); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4973, ANCOVA; Difference of adjusted means = -1.085, 95% CI 2-sided [-4.260 to 2.091], Standard Error of Mean 1.5889 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 3: Comparison: Placebo (R) vs 300 mg Lamotrigine (T1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0658, ANCOVA; Difference of adjusted means = -2.858, 95% CI 2-sided [-5.909 to 0.192], Standard Error of Mean 1.5266 — The difference was calculated as treatment group minus placebo group

3. Secondary Outcome: Rapid Visual Information Processing A' Prime (RVPA) on Ketamine
Description: Rapid Visual Information Processing (RVP) is a sensitive measure of sustained attention, outputting measures of response accuracy, target sensitivity and reaction times.
  The RVPA is a quantitative measure for a subject's sensitivity to the target sequence regardless of response tendency. The RVPA ranges from 0.00 to 1.00. The higher the RVPA value, the better the sensitivity to the target sequence one has.
Time Frame: At 4:20 and 5:06 hours:minutes after first drug administration in each treatment period.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- 25mg BI 425809 (T3): T3: 1 film-coated tablet of 25 milligrams (mg) BI 425809 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T3, 5 hours prior to ketamine infusion.
- 50mg BI 409306 (T2): T2: 1 film-coated tablet of 50 milligrams (mg) BI 409306 was administered orally once daily with 240 mL of water after a light snack on Day 1 of treatment T2, 2 hours prior to ketamine infusion.
- 300 mg Lamotrigine (T1): T1: 3 tablets of 100 milligrams (mg) Lamotrigine were administered orally once daily (daily dose: 300 mg) with 240 mL of water after a light snack on Day 1 of treatment T1, 2 hours prior to ketamine infusion.
Arm/Group | Placebo (R) | 25mg BI 425809 (T3) | 50mg BI 409306 (T2) | 300 mg Lamotrigine (T1)
Number analyzed (Participants) | 34 | 23 | 23 | 26
Score on a scale | 0.8743 (0.00702) | 0.8796 (0.00807) | 0.8800 (0.00810) | 0.9075 (0.00782)
Statistical Analysis 1: Comparison: Placebo (R) vs 25mg BI 425809 (T3); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.5081, ANCOVA; Difference of adjusted means = 0.0053, 95% CI 2-sided [-0.0106 to 0.0213], Standard Error of Mean 0.00798 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 2: Comparison: Placebo (R) vs 50mg BI 409306 (T2); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4723, ANCOVA; Difference of adjusted means = 0.0058, 95% CI 2-sided [-0.0102 to 0.0217], Standard Error of Mean 0.00798 — The difference was calculated as treatment group minus placebo group
Statistical Analysis 3: Comparison: Placebo (R) vs 300 mg Lamotrigine (T1); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < .0001, ANCOVA; Difference of adjusted means = 0.0333, 95% CI 2-sided [0.0180 to 0.0486], Standard Error of Mean 0.00767 — The difference was calculated as treatment group minus placebo group

ADVERSE EVENTS:
Time Frame: From intake of first study drug (00:00h planned time) up to Day 11 (03:00h planned time); Residual Effect Period (REP) of 11 days was used for each study treatment.
Description: Treated Set: The treated set included all subjects who were randomised and treated with at least one dose of Investigational medicinal product (IMP)/Placebo or ketamine.
Arm/Group | Placebo (R) | 25mg BI 425809 (T3) | 50mg BI 409306 (T2) | 300 mg Lamotrigine (T1)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/24 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/24 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 10/37 | 5/24 | 5/25 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (R) (N=37) | 25mg BI 425809 (T3) (N=24) | 50mg BI 409306 (T2) (N=25) | 300 mg Lamotrigine (T1) (N=26)
Nausea (Gastrointestinal disorders) | 2 | 4 | 4 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 1 | 0 | 1
Euphoric mood (Psychiatric disorders) | 3 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04602221/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04602221/SAP_001.pdf